CLINICAL TRIAL: NCT03046784
Title: Non-invasive Haemodynamic Monitoring in Pregnancy : Comparison Between Ultrasound and Nexfin Technology
Brief Title: Non-invasive Haemodynamic Monitoring in Pregnancy
Status: Completed | Type: Observational
Sponsor: Hospital Nord (Other)
Responsible Party: Principal Investigator, marc LEONE, Study Director, Clinical Professor, Hospital Nord
Other Study IDs: darnord2017-01
Record Dates: First submitted 2017-01-27; First posted 2017-02-08 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pregnancy Related; Cardiac Output, High; Haemodynamic Instability
MeSH Terms: conditions — Cardiac Output, High

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women in third trimester: Non-labouring pregnant women hospitalised during their third trimester of pregnancy has an haemodynamic evaluation with Nexfin technology and transthoracic cardiac ultrasonography.
  Evaluation is performed in two positions : dorsal decubitus and left lateral decubitus.
  Interventions: Other: haemodynamic evaluation

INTERVENTIONS:
Other: haemodynamic evaluation — continous haemodynamic monitoring is performed with digital Nexfin captor in two positions. in the same time transthoracic cardiac ultrasonography is performed to calculate cardiac output using velocity time index of aortic outflow chamber.

SUMMARY:
This prospective and observational trial over 55 pregnant women (third trimester) compares non invasive haemodynamic monitoring using Nexfin technology and ultrasonography technic

ELIGIBILITY:
Inclusion Criteria:

* third trimester of pregnancy
* Non-labouring pregnant women
* accepting study

Exclusion Criteria:

* refusal of study
* first or second trimester of pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregmant women
Study Population: Non-labouring term pregmant women in their third trimester
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiac output measure | 30 minutes
  Cardiac output is measured with non-invasive digital Nexfin technology (ml/min) and compared with transthoracic echocardiographic measure of cardiac output (ml/min) used as reference.
  Echographic cardiac output (ml/min) is measured as the produce of cross sectional aera of left ventricular outflow track (cm²) multiplied by velocity time index (cm) multiplied by heart rate (beat/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Departement anesthesie reanimation hopital nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montenij LJ, Buhre WF, Jansen JR, Kruitwagen CL, de Waal EE. Methodology of method comparison studies evaluating the validity of cardiac output monitors: a stepwise approach and checklist. Br J Anaesth. 2016 Jun;116(6):750-8. doi: 10.1093/bja/aew094. PMID 27199309
- [Background] Lee SW, Khaw KS, Ngan Kee WD, Leung TY, Critchley LA. Haemodynamic effects from aortocaval compression at different angles of lateral tilt in non-labouring term pregnant women. Br J Anaesth. 2012 Dec;109(6):950-6. doi: 10.1093/bja/aes349. Epub 2012 Oct 11. PMID 23059960